CLINICAL TRIAL: NCT03416933
Title: Therapeutic Drug Monitoring of Kinase Inhibitors and Study of Circulating Tumor DNA in Patients With Mutated BRAF Metastatic Cutaneous Melanoma and Treated With Anti-BRAF and Anti-MEK Kinase Inhibitors
Brief Title: Therapeutic Drug Monitoring of BRAF-mutated Advanced Melanoma
Acronym: OPTIMEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-A00469-46
Record Dates: First submitted 2018-01-18; First posted 2018-01-31 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Melanoma (Skin)
Keywords: ctDNA; MAPK inhibition; BRAF(V600) mutated
MeSH Terms: conditions — Melanoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological (Experimental)
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — 2x10 ml of patient peripherical blood will be collected at D0, D15, D30, D90, D180, D270 and with progression or at the end of the follow-up at the 12th month.

SUMMARY:
BRAF V600-mutant metastatic melanoma are commonly treated using a combination of anti-BRAF and anti-MEK tyrosine kinase inhibitors (TKIs). The OPTIMEL trial aims to study the interest of therapeutic drug monitoring (TDM) of TKIs and circulating tumor DNA (ctDNA) detected in plasma of patients with metastatic melanoma for disease monitoring. 35 patients with metastatic melanoma and treated with dabrafenib and trametinib will be enrolled in this trial. Blood samples will be collected for the determination of TKIs concentration and ctDNA detection.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years of age and older
* Histologic proven advanced skin melanoma (Stage IV or stage IIIc inoperable) with BRAF V600 mutation
* Patient who will treated with combined kinase inhibitors (dabrafenib + trametinib).
* Patient able to stand a blood collection of 20 mL
* Ability to provide an informed written consent form
* Patient must be affiliated to a social security system
* Patient's legal capacity to consent to study participation and to understand and comply with the requirements of the study.

Exclusion Criteria:

* Patient with mucosal melanoma
* Patient with non-metastatic skin melanoma (All stages except stage IV and stage III C inoperable)
* Patient with another synchronous cancer, or within 3 years
* Patient with a contraindication to blood collection of 20 mL
* Patient deprived of liberty or under supervision
* Patient unable to receive kinase inhibitor therapy
* Patient treated with another combined kinase inhibitors than dabrafenib and trametinib
* Pregnant or breastfeeding women
* Patient (man or woman) of childbearing age who does not agree to use of contraceptive methods validated during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Link between the presence of circulating tumor DNA and plasma concentrations of kinase inhibitors n patient with advanced BRAF(V600) mutated melanoma | 1 day
  ctDNA in patient with advanced BRAF(V600) mutated melanoma is estimated by the ratio of the Ct of the sample to the control. Plasma concentrations of anti-BRAF and anti-MEK tyrosine kinase inhibitors are expressed in μg / mL

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrois Lionnel, MD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (4):
- France (4):
  - Centre Georges François Leclerc (CGFL), Dijon
  - Hôpital de Mercy, Thionville
  - CHRU Nancy, Vandœuvre-lès-Nancy
  - Institut de Cancérologie de Lorraine (ICL), Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No